CLINICAL TRIAL: NCT02380547
Title: Sonographic Evaluation of Diaphragmatic Function in Critical Care Patients With Use of Non Invasive Ventilation
Acronym: ECHODIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5957
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Critical Care; Invasive Mechanical Ventilation
Keywords: Sonography; Diaphragmatic function; Non invasive ventilation; Critical care patients; Extubation after 24 hours of invasive ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Sonographic diaphragmatic measurements
  Other Names: Diaphragmatic excursion; Diaphragmatic thickening

SUMMARY:
Usefulness of non invasive ventilation in patients extubated after more than 48 hours of invasive ventilation is still in debate except for specific patients (chronic pulmonary disease and chronic heart failure).

Many experimental and clinical studies have shown that diaphragmatic function is depressed by mechanical ventilation in intubated patients.

The investigators will test the hypothesis that non invasive ventilation after extubation may improve diaphragmatic function

ELIGIBILITY:
Inclusion Criteria:

* Patient extubated after at least 48 hours of invasive ventilation
* Requiring non invasive ventilation
* Consent of patient

Exclusion Criteria:

* Diaphragmatic paralysis
* Neuromuscular disease
* significant pleural effusion
* atelectasis requiring bronchoscopy
* abdominal hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care patients (surgical or medical)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic excursion | Before the first NIV session
Diaphragmatic thickening | Before the first NIV session
Diaphragmatic excursion | After the first NIV session
Diaphragmatic thickening | After the first NIV session
Diaphragmatic excursion | After 24 h of NIV use
Diaphragmatic thickening | After 24 h of NIV use

CONTACTS AND LOCATIONS:
Overall Officials: Gharib AJOB, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service d'anesthésie- réanimation chirurgicale, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France